CLINICAL TRIAL: NCT02961972
Title: Effects of Oral Supplementation With Creatine on Plasma Homocysteine Levels and Systemic Microvascular Endothelial Function in Vegetarian Individuals
Brief Title: Effects of Oral Supplementation With Creatine on Systemic Microvascular Endothelial Function in Vegetarian Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Cardiology, Laranjeiras, Brazil (Other Government)
Responsible Party: Principal Investigator, Eduardo Tibirica, MD, PhD, National Institute of Cardiology, Laranjeiras, Brazil
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAAE: 302471512.4.0000.5272
Record Dates: First submitted 2016-11-07; First posted 2016-11-11 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Endothelial Dysfunction; Hyperhomocysteinemia
Keywords: vegetarianism; Hyperhomocysteinemia; vegan vegetarian
MeSH Terms: conditions — Hyperhomocysteinemia

STUDY DESIGN:
Intervention Model Description: creatine or placebo supplementation
Who Masked: Participant
Masking Description: creatine or placebo supplementation
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (Placebo Comparator): Oral ingestion of placebo pills (maltodextrin) during three weeks
  Interventions: Other: placebo
- creatine supplementation (Experimental): Oral supplementation with 5 g of monohydrate and micronized creatine during three weeks
  Interventions: Dietary Supplement: monohydrate and micronized creatine

INTERVENTIONS:
Dietary Supplement: monohydrate and micronized creatine — oral supplementation with creatine
  Arms: creatine supplementation
Other: placebo — oral supplementation with maltodextrin (control group)
  Arms: control group

SUMMARY:
The present study aims at investigating the effects of the oral supplementation with creatine on the systemic microvascular reactivity and plasma levels of homocysteine in vegetarian individuals of the vegan type.

DETAILED DESCRIPTION:
A vegetarian is an individual who lives on a diet of grains, pulses, legumes, nuts, seeds, vegetables, fruits, fungi, algae, yeast and/or some other non-animal-based foods, with or without, dairy products, honey and/or eggs. A vegetarian does not eat foods that consist of, or have been produced with the aid of products consisting of or created from, any part of the body of a living or dead animal. This includes meat, poultry, fish, shellfish, insects, by-products of slaughter** or any food made with processing aids created from these.

There are different types of vegetarian: i) Lacto-ovo-vegetarians eat both dairy products and eggs; this is the most common type of vegetarian diet; ii) Lacto-vegetarians eat dairy products but avoid eggs; iii) Ovo-vegetarians eat eggs but not dairy products; iv) Vegans do not eat dairy products, eggs, or any other products which are derived from animals.

Vegetarian individuals are considered to have lower cardiovascular risk for the development of cardiovascular diseases and lower cardiovascular mortality, when compared to omnivore individuals.

Nevertheless, some vegetarian diets may result in the deficiency of micronutrients and induce deficiency in some compounds such as vitamins, amino-acids, iron, zinc, calcium, omega-3 fatty acids and so on.

Moreover, vegetarian individuals can present deficiency in amino-acids such as carnosine and creatine, present essentially in the skeletal muscle of animals. In this context, deficiency in creatine has been considered as a risk factor for hyperhomocysteinemia and the consequent dysfunction of the vascular endothelium.

Hyperhomocysteinemia also is known to be an independent risk factor for cardiovascular diseases similar to hypertension, smoke and dyslipidemia.

In the present study, we investigate the effects of creatine supplementation in the systemic microvascular endothelial function and density in vegan-vegetarians presenting with normo- or hyperhomocysteinemia using laser-based skin flowmetry and video-capillaroscopy. We also investigate the effects of creatine supplementation on lipid and glycemic profile and plasma homocysteine levels.

Microvascular reactivity is evaluated using a laser speckle contrast imaging system in combination with the iontophoresis of acetylcholine (ACh), for the noninvasive and continuous measurement of cutaneous microvascular perfusion changes.

Microvascular density in the skin is evaluated using intravital video-microscopy.

ELIGIBILITY:
Inclusion Criteria:

* healthy vegetarians of the vegan type

Exclusion Criteria:

* previous treatment with dietary supplements
* high intensity physical activity

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2015-01; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Reactivity of the systemic microcirculation | three-week treatment
  Assessment of the endothelial-dependent microvascular reactivity in the skin using laser speckle contrast imaging

SECONDARY OUTCOMES:
cutaneous microvascular density | three-week treatment
  Assessment of skin microvascular density using video-capillaroscopy
Homocysteine levels in the plasma | three-week treatment

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Tibirica, MD, PhD, Principal Investigator — National Institute of Cardiology
Locations (1):
- National Institute of Cardiology, Ministry of Health, Brazil, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No